CLINICAL TRIAL: NCT00169182
Title: Randomized Study Comparing Induction Chemotherapy With Docetaxel, Cisplatin, 5FU Versus Cisplatin, 5 FU in Patients With T3 and T4 Larynx and Hypopharynx Carcinoma
Brief Title: Induction CT by Cisplatin, 5FU With or Without Docetaxel in Patients With T3 and T4 Larynx and Hypopharynx Carcinoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Groupe Oncologie Radiotherapie Tete et Cou (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GORTEC 2000-01
Record Dates: First submitted 2005-09-09; First posted 2005-09-15 (Estimated); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Larynx Cancer; Hypopharynx Cancer
Keywords: Larynx cancer; Hypopharynx cancer; Chemotherapy; Randomized trial; Larynx preservation
MeSH Terms: conditions — Laryngeal Neoplasms; Hypopharyngeal Neoplasms | interventions — Docetaxel; Cisplatin; 5-fluoro-3-pyridinecarboxylic acid

ARMS (2):
- TPF (Experimental): Docetaxel, Cisplatine, 5-FU
  Interventions: Drug: DOCETAXEL; Drug: Cisplatin; Drug: 5-Fluoro-3-Pyridinecarboxylic Acid
- PF (Active Comparator): Cisplatine, 5-FU
  Interventions: Drug: Cisplatin; Drug: 5-Fluoro-3-Pyridinecarboxylic Acid

INTERVENTIONS:
Drug: DOCETAXEL — 75 mg/m 2 on day 1
  Arms: TPF
Drug: Cisplatin — 75 mg/m 2 on day 1
Drug: 5-Fluoro-3-Pyridinecarboxylic Acid — 750 mg/m 2 by 24-hour continuous infusion for 5 days

SUMMARY:
The purpose of the study is to compare two regimen of chemotherapy used as first treatment for patients with larynx or hypopharynx tumors that would be treated with total laryngectomy. The standard treatment is a combination of 2 drugs (Cisplatin and 5FU). The aim of the study is to evaluate the potential benefit of the addition of a third drug (Docetaxel) in the chemotherapy regimen. Patients will receive 3 cycles of chemotherapy. Responders to the induction treatment are treated with radiation with a purpose of larynx preservation. Non responders patients will be treated with total laryngectomy.

DETAILED DESCRIPTION:
The purpose of the study is to compare two regimen of induction chemotherapy for patients with T3 and T4 larynx or hypopharynx carcinoma that would be treated with total laryngectomy. The aim of the study is to compare the standard regimen (Cisplatin + 5FU) versus the TPF regimen (Taxotere + Cisplatin + 5FU). Responders to the induction treatment are treated with radiation with a purpose of larynx preservation. Non responders patients will be treated with total laryngectomy followed by postoperative radiation.

ELIGIBILITY:
Inclusion Criteria:

* T3 and T4 larynx and hypopharynx tumor that would be treated with total laryngectomy
* Biopsy proven carcinoma
* Adequate biology
* Performance status 0 or 1

Exclusion Criteria:

* Larynx or hypopharynx tumors that could be treated with partial laryngectomy
* Distant metastasis
* Prior surgery, chemotherapy or radiation
* Intercurrent disease that is a contra indication to chemotherapy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2001-12-15 (Actual); Primary Completion 2009-04 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
3-years larynx preservation rate

SECONDARY OUTCOMES:
5-years survival rate

CONTACTS AND LOCATIONS:
Overall Officials: Gilles Calais, MD, Principal Investigator — CHU Bretonneau
Locations (1):
- CHU Bretonneau, Tours, France